CLINICAL TRIAL: NCT03900325
Title: A Single-Blind Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Exploratory Efficacy of Nimacimab in Patients With Diabetic Gastroparesis
Brief Title: Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Exploratory Efficacy of Nimacimab in Patients With Diabetic Gastroparesis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Bird Rock Bio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: BRB-018-200DG
Record Dates: First submitted 2019-03-27; First posted 2019-04-03 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2019-08

CONDITIONS: Diabetic Gastroparesis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Nimacimab (Experimental): 2.5 mg/kg
  Interventions: Drug: Nimacimab
- Placebo (Placebo Comparator): 0.9% sodium chloride
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nimacimab — 2.5 mg/kg
  Arms: Nimacimab
Drug: Placebo — 0.9% sodium chloride
  Arms: Placebo

SUMMARY:
This is a single blind phase 2a study to evaluate the safety, tolerability, pharmacokinetics, and exploratory efficacy of nimacimab in patients with diabetic gastroparesis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with type 1 or type 2 diabetes
* Diagnosed with diabetic gastroparesis, defined by:

  1. 3 month past or current history of symptoms of gastroparesis (e.g. nausea, vomiting, bloating, abdominal pain, or feeling full earlier than normal after eating)
  2. Screening or historical scintigraphy (3 years prior to screening) with > 20% of solid contents retained at 4 hours.
* BMI >= 20.0 and < = 50.0 kg/m2

Exclusion Criteria:

* Participants on prokinetic therapy should have these medications withdrawn at least 7 days prior to any study scintigraphy exam and at least 7 days prior to the first dose through Day 15 of treatment.
* Participants with any active prokinetic device are excluded, unless device is turned off for at least 7 days prior to any study scintigraphy exam and at least 7 days prior to the first dose through Day 15 of treatment.
* Participants who are currently participating in or have participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study intervention.
* Participants with uncontrolled diabetes. Participants with controlled diabetes are allowed (insulin is allowed). HbA1c>9.9% at screening are excluded.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-01 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
Frequency of clinically significant laboratory abnormalities | Day 38
Frequency of clinically significant vital signs | Day 38
Frequency of clinically significant ECGs | Day 38

SECONDARY OUTCOMES:
Nimacimab serum concentration | Day 3, Day 8, Day 10, Day 38
  Area under the plasma concentration versus time curve (AUC)

OTHER OUTCOMES:
Measure rate of gastric emptying after ingestion of a radio-labeled meal as measured by gamma scans (scintigraphy) at 0, 0.5, 1, 2, 3, and 4 hours post meal | Baseline, Day 10
Gastric emptying half-time as measured by gamma scans (scintigraphy) after ingestion of a radio-labeled meal. | Baseline, Day 10
  Half time (t1/2) of gastric emptying (GE) of solids is the time for half of the ingested solids or liquids to leave the stomach.
Change from baseline in American Neurogastroenterology and Motility Society Gastroparesis Cardinal Symptom Index Daily Diary (GCSI-DD) Composite Score at 15 days | Baseline and 15 days
  The ANMS GCSI-DD composite score includes score of nausea, early satiety, upper abdominal pain and postprandial fullness. The severity scores of these symptoms range from 0 ( none) to 4 (very severe).

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Panax Clinical Research, Miami, Florida
  - International Research Associates, LLC, Miami, Florida
  - PRN of Kansas, Wichita, Kansas
  - Mayo Clinic, Rochester, Minnesota
  - ClinSearch, Chattanooga, Tennessee